CLINICAL TRIAL: NCT06289257
Title: Analysis of Vitamin D and VDR Expression in Women With Advanced Endometriosis: A Case-Control Study in Thailand
Brief Title: Analysis of Vitamin D and VDR Expression in Endometriosis: A Case-Control Study
Status: Completed | Type: Observational
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Vitet Layanun, Dr.Vitet Layanun, Khon Kaen University
Other Study IDs: HE661574
Record Dates: First submitted 2024-02-20; First posted 2024-03-01 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Endometriosis; Vitamin D Deficiency/Insufficiency; Vitamin D Status
Keywords: Vitamin D level; Endometriosis; Vitamin D receptor; rASRM; Immunohistochemistry; 25(OH)D
MeSH Terms: conditions — Endometriosis; Vitamin D Deficiency | interventions — Receptors, Calcitriol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood for Vitamin D level<25(OH)D, Calcium, Phosphate, Magnesium, Albumin, AST, ALT, Creatinine, Tissue for Anti VDR staining.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Endometriosis: Women with endometriosis
  Interventions: Diagnostic Test: Vitamin D level; Other: Vitamin D receptor
- Control: Healthy women
  Interventions: Diagnostic Test: Vitamin D level

INTERVENTIONS:
Diagnostic Test: Vitamin D level — Vitamin D level in blood
  Other Names: Vitamin D status
Other: Vitamin D receptor — Vitamin D receptor in endometriosis tissue
  Groups: Endometriosis

SUMMARY:
The goal of this cross-sectional prospective matching study is to evaluate whether serum vitamin D levels and vitamin D receptor (VDR) expression are associated with the presence and severity of endometriosis in women of reproductive age.

The main questions it aims to answer are:

* Is there a difference in serum 25-hydroxyvitamin D [25(OH)D] levels between women with endometriosis and healthy controls?
* Is there a correlation between serum vitamin D levels and VDR expression in endometriotic tissues?
* Is there an association between vitamin D status and the severity of endometriosis based on the revised American Society for Reproductive Medicine (rASRM) staging?

Researchers will compare participants with endometriosis to matched healthy controls (1:2 ratio).

Participants will:

* Provide blood samples for serum 25(OH)D measurement.
* Undergo surgical tissue sampling (for the endometriosis group) to assess VDR expression using immunohistochemistry staining.
* Complete structured questionnaires regarding sun exposure, lifestyle, and clinical characteristics.

DETAILED DESCRIPTION:
This cross-sectional study aims to investigate the association between serum vitamin D levels and endometriosis, and to further explore the expression of vitamin D receptor (VDR) in endometriotic tissues using immunohistochemistry.

The study enrolled reproductive-aged women diagnosed with endometriosis who underwent laparoscopic surgery and compared them with matched healthy controls based on age and BMI.

Serum levels of 25-hydroxyvitamin D [25(OH)D] were measured using a standardized laboratory assay. Endometriotic tissue samples obtained during surgery were analyzed for VDR expression, qualitative-quantified using the H-score method in both stroma and epithelial compartments. Clinical data, including revised American Society for Reproductive Medicine (rASRM) staging, were used to assess disease severity. Additional data were collected via structured interviews covering sun exposure, reproductive history, lifestyle, and hormonal treatment.

Tissue staining and scoring were reviewed by two blinded pathologists to ensure reproducibility. Data entry validation was performed by cross-checking case report forms with original clinical records, and double data entry methods were used to minimize errors.

Sample size was determined based on prior effect size estimates from published literature, aiming to achieve a power of 80% and significance level of 5%. The study population was sufficient to detect a clinically meaningful difference in vitamin D status between cases and controls.

Missing data were managed using complete case analysis and sensitivity checks. For secondary outcomes, subgroup analyses were conducted based on categorized vitamin D levels (normal, insufficiency, deficiency, severe deficiency).

Statistical analysis included:

* Descriptive statistics for demographic and clinical characteristics.
* Conditional logistic regression or non-parametric equivalents for between-group comparisons.
* Logistic regression models to estimate the odds ratios for severe endometriosis by vitamin D status.
* Correlation analyses between serum vitamin D levels, VDR expression (H-scores), and rASRM scores.

All analyses were performed using STATA version 18.5. The findings aim to clarify the potential role of vitamin D and its receptor in endometriosis pathogenesis and to inform future interventional studies and clinical practice.

ELIGIBILITY:
Inclusion Criteria Endometriosis Group:

* Women diagnosed with ectopic endometriotic tissue:
* Have a scheduled surgery appointment at Sri Nakarin Hospital.
* Are aged 18 years or older.

Inclusion Criteria Control Group:

* Women undergoing examination at the outpatient department of Sri Nakarin Hospital.
* No history of gynecological diseases or previous treatment for gynecological conditions associated with lower abdominal pain, infections, or abdominal masses at present.
* Have undergone a gynecological examination within the past year, or if examined during the current visit, the results were normal.
* Have undergone an ultrasound examination within the past year, or if examined during the current visit, the ultrasound results were normal.

Exclusion Criteria:

* Received vitamin D supplements within the past 3 months prior to volunteering.
* History of chronic infectious diseases.
* Previously treated for autoimmune diseases.
* History of polycystic ovarian.
* History of bone disorders or receiving medications affecting bones.
* Irregular menstrual cycles or absence of menstruation for more than 3 months up to 1 year.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thai women, reproductive age
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Vitamin D level | At enrollment
  Vitamin D status

SECONDARY OUTCOMES:
rASRM | Intra operation
  Severity of the disease
Vitamin D receptor | Up to 4 weeks after surgery
  Tissue staining of Vitamin D antibody

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Faculty of Medicine, Khonkaen University, Khon Kaen, Changwat Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No
Follow the Center for Ethics in Human Research, Khon Kaen University submission.

REFERENCES:
- [Background] Pludowski P, Takacs I, Boyanov M, Belaya Z, Diaconu CC, Mokhort T, Zherdova N, Rasa I, Payer J, Pilz S. Clinical Practice in the Prevention, Diagnosis and Treatment of Vitamin D Deficiency: A Central and Eastern European Expert Consensus Statement. Nutrients. 2022 Apr 2;14(7):1483. doi: 10.3390/nu14071483. PMID 35406098
- [Background] Anglesio MS, Papadopoulos N, Ayhan A, Nazeran TM, Noe M, Horlings HM, Lum A, Jones S, Senz J, Seckin T, Ho J, Wu RC, Lac V, Ogawa H, Tessier-Cloutier B, Alhassan R, Wang A, Wang Y, Cohen JD, Wong F, Hasanovic A, Orr N, Zhang M, Popoli M, McMahon W, Wood LD, Mattox A, Allaire C, Segars J, Williams C, Tomasetti C, Boyd N, Kinzler KW, Gilks CB, Diaz L, Wang TL, Vogelstein B, Yong PJ, Huntsman DG, Shih IM. Cancer-Associated Mutations in Endometriosis without Cancer. N Engl J Med. 2017 May 11;376(19):1835-1848. doi: 10.1056/NEJMoa1614814. PMID 28489996
- [Background] Sampson JA. Peritoneal endometriosis due to the menstrual dissemination of endometrial tissue into the peritoneal cavity. American Journal of Obstetrics and Gynecology. 1927;14(4):422-69.
- [Background] Yu K, Huang ZY, Xu XL, Li J, Fu XW, Deng SL. Estrogen Receptor Function: Impact on the Human Endometrium. Front Endocrinol (Lausanne). 2022 Feb 28;13:827724. doi: 10.3389/fendo.2022.827724. eCollection 2022. PMID 35295981
- [Background] Agic A, Xu H, Altgassen C, Noack F, Wolfler MM, Diedrich K, Friedrich M, Taylor RN, Hornung D. Relative expression of 1,25-dihydroxyvitamin D3 receptor, vitamin D 1 alpha-hydroxylase, vitamin D 24-hydroxylase, and vitamin D 25-hydroxylase in endometriosis and gynecologic cancers. Reprod Sci. 2007 Jul;14(5):486-97. doi: 10.1177/1933719107304565. PMID 17913968
- [Background] Bulun SE. Yen and Jaffe's Reproductive Endocrinology: Physiology, Pathophysiology and Clinical Management, 9th edition. 9 ed: Elsevier; 2023 12/07/2023. 1040 p.
- [Background] Bulun SE, Yilmaz BD, Sison C, Miyazaki K, Bernardi L, Liu S, Kohlmeier A, Yin P, Milad M, Wei J. Endometriosis. Endocr Rev. 2019 Aug 1;40(4):1048-1079. doi: 10.1210/er.2018-00242. PMID 30994890
- [Background] Bulun SE, Yildiz S, Adli M, Chakravarti D, Parker JB, Milad M, Yang L, Chaudhari A, Tsai S, Wei JJ, Yin P. Endometriosis and adenomyosis: shared pathophysiology. Fertil Steril. 2023 May;119(5):746-750. doi: 10.1016/j.fertnstert.2023.03.006. Epub 2023 Mar 15. PMID 36925057
- [Background] Suda K, Nakaoka H, Yoshihara K, Ishiguro T, Tamura R, Mori Y, Yamawaki K, Adachi S, Takahashi T, Kase H, Tanaka K, Yamamoto T, Motoyama T, Inoue I, Enomoto T. Clonal Expansion and Diversification of Cancer-Associated Mutations in Endometriosis and Normal Endometrium. Cell Rep. 2018 Aug 14;24(7):1777-1789. doi: 10.1016/j.celrep.2018.07.037. PMID 30110635
- [Background] Inoue S, Hirota Y, Ueno T, Fukui Y, Yoshida E, Hayashi T, Kojima S, Takeyama R, Hashimoto T, Kiyono T, Ikemura M, Taguchi A, Tanaka T, Tanaka Y, Sakata S, Takeuchi K, Muraoka A, Osuka S, Saito T, Oda K, Osuga Y, Terao Y, Kawazu M, Mano H. Uterine adenomyosis is an oligoclonal disorder associated with KRAS mutations. Nat Commun. 2019 Dec 19;10(1):5785. doi: 10.1038/s41467-019-13708-y. PMID 31857578
- [Background] Lips P. Vitamin D physiology. Prog Biophys Mol Biol. 2006 Sep;92(1):4-8. doi: 10.1016/j.pbiomolbio.2006.02.016. Epub 2006 Feb 28. PMID 16563471
- [Background] Wimalawansa SJ. Infections and Autoimmunity-The Immune System and Vitamin D: A Systematic Review. Nutrients. 2023 Sep 2;15(17):3842. doi: 10.3390/nu15173842. PMID 37686873
- [Background] Chailurkit LO, Aekplakorn W, Ongphiphadhanakul B. Regional variation and determinants of vitamin D status in sunshine-abundant Thailand. BMC Public Health. 2011 Nov 10;11:853. doi: 10.1186/1471-2458-11-853. PMID 22074319
- [Background] Rajatanavin N, Kanokrungsee S, Aekplakorn W. Vitamin D status in Thai dermatologists and working-age Thai population. J Dermatol. 2019 Mar;46(3):206-212. doi: 10.1111/1346-8138.14742. Epub 2018 Dec 28. PMID 30592077
- [Background] Jiang Z, Pu R, Li N, Chen C, Li J, Dai W, Wang Y, Hu J, Zhu D, Yu Q, Shi Y, Yang G. High prevalence of vitamin D deficiency in Asia: A systematic review and meta-analysis. Crit Rev Food Sci Nutr. 2023;63(19):3602-3611. doi: 10.1080/10408398.2021.1990850. Epub 2021 Nov 16. PMID 34783278
- [Background] Cashman KD. Global differences in vitamin D status and dietary intake: a review of the data. Endocr Connect. 2022 Jan 11;11(1):e210282. doi: 10.1530/EC-21-0282. PMID 34860171
- [Background] Md Isa Z, Mohd Nordin NR, Mahmud MH, Hashim S. An Update on Vitamin D Deficiency Status in Malaysia. Nutrients. 2022 Jan 27;14(3):567. doi: 10.3390/nu14030567. PMID 35276926
- [Background] Tuyen le D, Hien VT, Binh PT, Yamamoto S. Calcium and Vitamin D Deficiency in Vietnamese: Recommendations for an Intervention Strategy. J Nutr Sci Vitaminol (Tokyo). 2016;62(1):1-5. doi: 10.3177/jnsv.62.1. PMID 27117844
- [Background] Pludowski P. Supplementing Vitamin D in Different Patient Groups to Reduce Deficiency. Nutrients. 2023 Aug 25;15(17):3725. doi: 10.3390/nu15173725. PMID 37686757
- [Background] Horikawa A, Kasukawa Y, Hongo M, Kodama H, Sano A, Miyakoshi N. A prospective analysis of concentration of 25-OHD between northern and southern district in Japan in year-round study. Medicine (Baltimore). 2022 Oct 28;101(43):e31340. doi: 10.1097/MD.0000000000031340. PMID 36316947
- [Background] Hartwell D, Rodbro P, Jensen SB, Thomsen K, Christiansen C. Vitamin D metabolites--relation to age, menopause and endometriosis. Scand J Clin Lab Invest. 1990 Apr;50(2):115-21. doi: 10.3109/00365519009089142. PMID 2339276
- [Background] Neale RE, Khan SR, Lucas RM, Waterhouse M, Whiteman DC, Olsen CM. The effect of sunscreen on vitamin D: a review. Br J Dermatol. 2019 Nov;181(5):907-915. doi: 10.1111/bjd.17980. Epub 2019 Jul 9. PMID 30945275
- [Background] Martelli M, Salvio G, Santarelli L, Bracci M. Shift Work and Serum Vitamin D Levels: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2022 Jul 22;19(15):8919. doi: 10.3390/ijerph19158919. PMID 35897284
- [Background] Walsh JS, Bowles S, Evans AL. Vitamin D in obesity. Curr Opin Endocrinol Diabetes Obes. 2017 Dec;24(6):389-394. doi: 10.1097/MED.0000000000000371. PMID 28915134
- [Background] Zakharova I, Klimov L, Kuryaninova V, Nikitina I, Malyavskaya S, Dolbnya S, Kasyanova A, Atanesyan R, Stoyan M, Todieva A, Kostrova G, Lebedev A. Vitamin D Insufficiency in Overweight and Obese Children and Adolescents. Front Endocrinol (Lausanne). 2019 Mar 1;10:103. doi: 10.3389/fendo.2019.00103. eCollection 2019. PMID 30881343
- [Background] Karampela I, Sakelliou A, Vallianou N, Christodoulatos GS, Magkos F, Dalamaga M. Vitamin D and Obesity: Current Evidence and Controversies. Curr Obes Rep. 2021 Jun;10(2):162-180. doi: 10.1007/s13679-021-00433-1. Epub 2021 Apr 1. PMID 33792853
- [Background] Huang X, Yang Y, Jiang Y, Zhou Z, Zhang J. Association between vitamin D deficiency and lipid profiles in overweight and obese adults: a systematic review and meta-analysis. BMC Public Health. 2023 Aug 29;23(1):1653. doi: 10.1186/s12889-023-16447-4. PMID 37644450
- [Background] Wang H, Chen W, Li D, Yin X, Zhang X, Olsen N, Zheng SG. Vitamin D and Chronic Diseases. Aging Dis. 2017 May 2;8(3):346-353. doi: 10.14336/AD.2016.1021. eCollection 2017 May. PMID 28580189
- [Background] Halder SK, Osteen KG, Al-Hendy A. Vitamin D3 inhibits expression and activities of matrix metalloproteinase-2 and -9 in human uterine fibroid cells. Hum Reprod. 2013 Sep;28(9):2407-16. doi: 10.1093/humrep/det265. Epub 2013 Jun 27. PMID 23814095
- [Background] Kure S, Nosho K, Baba Y, Irahara N, Shima K, Ng K, Meyerhardt JA, Giovannucci EL, Fuchs CS, Ogino S. Vitamin D receptor expression is associated with PIK3CA and KRAS mutations in colorectal cancer. Cancer Epidemiol Biomarkers Prev. 2009 Oct;18(10):2765-72. doi: 10.1158/1055-9965.EPI-09-0490. Epub 2009 Sep 29. PMID 19789368
- [Background] Matasariu DR, Mandici CE, Ursache A, Bausic AIG, Bujor IE, Cristofor AE, Boiculese LV, Grigore M, Bratila E, Lozneanu L. Vitamin D and Mitosis Evaluation in Endometriosis: A Step toward Discovering the Connection? Biomedicines. 2023 Jul 26;11(8):2102. doi: 10.3390/biomedicines11082102. PMID 37626598
- [Background] Miyashita M, Koga K, Izumi G, Sue F, Makabe T, Taguchi A, Nagai M, Urata Y, Takamura M, Harada M, Hirata T, Hirota Y, Wada-Hiraike O, Fujii T, Osuga Y. Effects of 1,25-Dihydroxy Vitamin D3 on Endometriosis. J Clin Endocrinol Metab. 2016 Jun;101(6):2371-9. doi: 10.1210/jc.2016-1515. Epub 2016 Apr 1. PMID 27035829
- [Background] Krishnan AV, Swami S, Feldman D. The potential therapeutic benefits of vitamin D in the treatment of estrogen receptor positive breast cancer. Steroids. 2012 Sep;77(11):1107-12. doi: 10.1016/j.steroids.2012.06.005. Epub 2012 Jul 16. PMID 22801352
- [Background] Matsuzaki S, Murakami T, Uehara S, Canis M, Sasano H, Okamura K. Expression of estrogen receptor alpha and beta in peritoneal and ovarian endometriosis. Fertil Steril. 2001 Jun;75(6):1198-205. doi: 10.1016/s0015-0282(01)01783-6. PMID 11384649
- [Background] Pluchino N, Mamillapalli R, Wenger JM, Ramyead L, Drakopoulos P, Tille JC, Taylor HS. Estrogen receptor-alpha immunoreactivity predicts symptom severity and pain recurrence in deep endometriosis. Fertil Steril. 2020 Jun;113(6):1224-1231.e1. doi: 10.1016/j.fertnstert.2020.01.036. Epub 2020 May 13. PMID 32416979
- [Background] Andersen CL, Boisen MM, Sikora MJ, Ma T, Tseng G, Suryawanshi S, Vlad A, Elishaev E, Edwards RP, Oesterreich S. The Evolution of Estrogen Receptor Signaling in the Progression of Endometriosis to Endometriosis-Associated Ovarian Cancer. Horm Cancer. 2018 Dec;9(6):399-407. doi: 10.1007/s12672-018-0350-9. Epub 2018 Oct 9. PMID 30302736
- [Background] Chantalat E, Valera MC, Vaysse C, Noirrit E, Rusidze M, Weyl A, Vergriete K, Buscail E, Lluel P, Fontaine C, Arnal JF, Lenfant F. Estrogen Receptors and Endometriosis. Int J Mol Sci. 2020 Apr 17;21(8):2815. doi: 10.3390/ijms21082815. PMID 32316608
- [Background] Becker CM, Bokor A, Heikinheimo O, Horne A, Jansen F, Kiesel L, King K, Kvaskoff M, Nap A, Petersen K, Saridogan E, Tomassetti C, van Hanegem N, Vulliemoz N, Vermeulen N; ESHRE Endometriosis Guideline Group. ESHRE guideline: endometriosis. Hum Reprod Open. 2022 Feb 26;2022(2):hoac009. doi: 10.1093/hropen/hoac009. eCollection 2022. PMID 35350465
- [Background] Revised American Society for Reproductive Medicine classification of endometriosis: 1996. Fertil Steril. 1997 May;67(5):817-21. doi: 10.1016/s0015-0282(97)81391-x. No abstract available. PMID 9130884
- [Background] Orr NL, Albert A, Liu YD, Lum A, Hong J, Ionescu CL, Senz J, Nazeran TM, Lee AF, Noga H, Lawrenson K, Allaire C, Williams C, Bedaiwy MA, Anglesio MS, Yong PJ. KRAS mutations and endometriosis burden of disease. J Pathol Clin Res. 2023 Jul;9(4):302-312. doi: 10.1002/cjp2.317. Epub 2023 Mar 28. PMID 36977195
- [Background] Ke J, Ye J, Li M, Zhu Z. The Role of Matrix Metalloproteinases in Endometriosis: A Potential Target. Biomolecules. 2021 Nov 22;11(11):1739. doi: 10.3390/biom11111739. PMID 34827737
- [Background] Ueda M, Yamashita Y, Takehara M, Terai Y, Kumagai K, Ueki K, Kanda K, Hung YC, Ueki M. Gene expression of adhesion molecules and matrix metalloproteinases in endometriosis. Gynecol Endocrinol. 2002 Oct;16(5):391-402. PMID 12587534
- [Background] Sharpe-Timms KL, Cox KE. Paracrine regulation of matrix metalloproteinase expression in endometriosis. Ann N Y Acad Sci. 2002 Mar;955:147-56; discussion 157-8, 396-406. doi: 10.1111/j.1749-6632.2002.tb02775.x. PMID 11949944
- [Background] MacLean JA 2nd, Hayashi K. Progesterone Actions and Resistance in Gynecological Disorders. Cells. 2022 Feb 13;11(4):647. doi: 10.3390/cells11040647. PMID 35203298
- [Background] Zhang P, Wang G. Progesterone Resistance in Endometriosis: Current Evidence and Putative Mechanisms. Int J Mol Sci. 2023 Apr 10;24(8):6992. doi: 10.3390/ijms24086992. PMID 37108154
- [Background] Zheng SH, Chen XX, Chen Y, Wu ZC, Chen XQ, Li XL. Antioxidant vitamins supplementation reduce endometriosis related pelvic pain in humans: a systematic review and meta-analysis. Reprod Biol Endocrinol. 2023 Aug 29;21(1):79. doi: 10.1186/s12958-023-01126-1. PMID 37644533
- [Background] Harris HR, Chavarro JE, Malspeis S, Willett WC, Missmer SA. Dairy-food, calcium, magnesium, and vitamin D intake and endometriosis: a prospective cohort study. Am J Epidemiol. 2013 Mar 1;177(5):420-30. doi: 10.1093/aje/kws247. Epub 2013 Feb 3. PMID 23380045
- [Background] Kahlon BK, Simon-Collins M, Nylander E, Segars J, Singh B. A systematic review of vitamin D and endometriosis: role in pathophysiology, diagnosis, treatment, and prevention. F&S Reviews. 2023;4(1):1-14.
- [Background] Delbandi AA, Torab M, Abdollahi E, Khodaverdi S, Rokhgireh S, Moradi Z, Heidari S, Mohammadi T. Vitamin D deficiency as a risk factor for endometriosis in Iranian women. J Reprod Immunol. 2021 Feb;143:103266. doi: 10.1016/j.jri.2020.103266. Epub 2020 Dec 17. PMID 33385732
- [Background] Denisova AS, Yarmolinskaya MI, Tkachenko NN. Assessment of 25(OH)D status in patients with genital endometriosis and clinical efficacy of cholecalciferol in the treatment of the disease. JOWD. 2021;70(4):125-33.
- [Background] Cho MC, Kim JH, Jung MH, Cho IA, Jo HC, Shin JK, Lee SA, Choi WJ, Lee JH. Analysis of vitamin D-binding protein (VDBP) gene polymorphisms in Korean women with and without endometriosis. Clin Exp Reprod Med. 2019 Sep;46(3):132-139. doi: 10.5653/cerm.2019.00122. Epub 2019 Aug 13. PMID 31405270
- [Background] Buggio L, Somigliana E, Pizzi MN, Dridi D, Roncella E, Vercellini P. 25-Hydroxyvitamin D Serum Levels and Endometriosis: Results of a Case-Control Study. Reprod Sci. 2019 Feb;26(2):172-177. doi: 10.1177/1933719118766259. Epub 2018 Mar 27. PMID 29587615
- [Background] Baek JC, Jo JY, Lee SM, Cho IA, Shin JK, Lee SA, Lee JH, Cho MC, Choi WJ. Differences in 25-hydroxy vitamin D and vitamin D-binding protein concentrations according to the severity of endometriosis. Clin Exp Reprod Med. 2019 Sep;46(3):125-131. doi: 10.5653/cerm.2018.00416. Epub 2019 Aug 1. PMID 31370113
- [Background] Anastasi E, Fuggetta E, De Vito C, Migliara G, Viggiani V, Manganaro L, Granato T, Benedetti Panici P, Angeloni A, Porpora MG. Low levels of 25-OH vitamin D in women with endometriosis and associated pelvic pain. Clin Chem Lab Med. 2017 Oct 26;55(12):e282-e284. doi: 10.1515/cclm-2017-0016. No abstract available. PMID 28453438
- [Background] Derakhshan M, Derakhshan M, Hedayat P, Shiasi M, Sadeghi E, editors. Vitamin D Deficiency May Be a Modifiable Risk Factor in Women With Endometriosis2018.
- [Background] Somigliana E, Panina-Bordignon P, Murone S, Di Lucia P, Vercellini P, Vigano P. Vitamin D reserve is higher in women with endometriosis. Hum Reprod. 2007 Aug;22(8):2273-8. doi: 10.1093/humrep/dem142. Epub 2007 Jun 4. PMID 17548365